CLINICAL TRIAL: NCT05512624
Title: Integrating an Evidence-based Mental Health Intervention Into Primary Health Care to Improve Outcomes for Refugees With Hypertension, Diabetes, and Epilepsy
Brief Title: Integrating a Mental Health Intervention Into Primary Health Care for Refugees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Rescue Committee (Other)
Collaborators: Khon Kaen University (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EX175
Record Dates: First submitted 2022-05-15; First posted 2022-08-23 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Medication Adherence; Mental Health Issue; Self Efficacy; Hypertension; Epilepsy; Diabetes
MeSH Terms: conditions — Medication Adherence; Hypertension; Epilepsy; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Two-armed randomized waitlisted control trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The course of Common Elements Treatment Approach (CETA - the intervention under study) is built to be flexible depending on need. Mild symptoms could result in fewer sessions (e.g., 5), while greater severity may require 8-12 sessions.
  Interventions: Behavioral: Common Elements Treatment Approach
- Waitlisted Arm (No Intervention): The waitlisted arm will be offered the CETA approach upon conclusion of the endline data collection.

INTERVENTIONS:
Behavioral: Common Elements Treatment Approach — For treatment group participants, they will then have weekly meetings with a counselor lasting no more than 1.5 hours per session, and a total of approximately 10 sessions. Both treatment and wait list participants will then complete the assessment instrument at 3 months and 6 months post-enrollment (each lasting no more than 1.5 hours). All total, it is expected that treatment group participants will have up to 13 meetings with a study team member or counselor over the course of their participation.
  Wait list group participants will have 3 meetings with a study team member over the course of their participation. If the treatment is deemed to be effective these wait list participants will be the first adults to be offered the intervention after trial completion.
  Arms: Intervention Arm

SUMMARY:
The objective of this study is to evaluate the impact of an evidence-based mental health intervention (Common Elements Treatment Approach) on medication adherence, behavioral improvement and clinical outcomesamong adults taking medication for hypertension, diabetes and epilepsy using a two-arm randomized wait-list controlled trial among adult refugees in Mae La camp, Thailand.

ELIGIBILITY:
Inclusion Criteria:

* A. Inclusion criteria:

  1. Patients who was diagnosed by physician based on ICD 10 to have diabetes, hypertension or diabetes with hypertension comorbidity, or epilepsy.
  2. Registered in chronic database system of the camp.

B. Exclusion criteria:

1. who are younger than 18 years old
2. who have severe physical illness
3. who have severe mental disorders
4. who will not stay in the camp until the end of the program
5. who are not willing to participate in the program

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence Report Scale | Baseline, Endline, Past two weeks
  Medication Adherence - Self Report will be assessed using the 5-item Medication Adherence Report Scale (MARS-5). Each item assesses the frequency of deviations in medication use, ranging from never (0) to all days (4) over the past two weeks. The MARS-5 will be scored by calculating the mean of all items to generate a continuous score ranging from 0-4, with higher scores indicating greater problems with medication adherence.
Pill Count Medication Adherence | Baseline, Endline, Past two weeks
  Medication Adherence - Pill Count: Measurement: Medication Adherence will also be objectively measured by counting the proportion of pills taken over the past two weeks relative to the number taken if used as prescribed over the same period. Proportions will range from 0-100% with higher proportion indicating greater adherence. Proportions will be used to classify a binary indicator of adherence using an 80% or higher cutoff.

OTHER OUTCOMES:
Substance use | Baseline, Endline, Past two weeks
  two locally developed items each assessing self-reported use of alcohol, tobacco, and betel nut. The first question for each substance assesses frequency of use, ranging from never (0) to all days (4) over the past two weeks. The second item is open-ended to record self-reported daily average intake (drinks/smokes/betels per day). Separate consumption scores will be generated for each of alcohol, tobacco, and betel by multiplying the frequency range (0-4) by the average intake to generate a continuous numeric quantifier of recent consumption, with higher scores reflecting greater consumption.
Physical activity | Baseline, Endline, Past two weeks
  Three locally developed items assessing frequency of physical activities (vigorous, moderate, and leisure) for at least 30 minutes, ranging from never (0) to all days (4) over the past two weeks. A composite score will be calculated by taking the mean of all 3 items , for a total score ranging from 0-4 with higher scores indicating greater frequency of physical activity.
Diet | Baseline, Endline, Past two weeks
  Three locally developed items assessing frequency of unhealthy food consumption (sugary, fatty, and salty foods), ranging from never (0) to all days (4) over the past two weeks. A composite score will be calculated by taking the mean of all 3 items, for a total score ranging from 0-4 with higher scores indicating greater consumption of unhealthy foods.
Sleep Quality | Baseline, Endline, Past two weeks
  Sleep quality will be assessed using the 6-item sleep scale from the Medical Outcomes Study (MOS-6). Items assess frequency of experiencing a range of positive (2 items) and problematic (4 items) sleep experiences, ranging from none of the time (0) to all of the time (4) over the past two weeks. The MOS-6 will be scored by first reverse-scoring the two positively worded items, then calculating the mean of all items to generate a continuous score ranging from 0-4, with higher scores indicating poorer sleep patterns.
Mental Health Symptoms | Baseline, Endline, Past two weeks
  The Myanmar-Wide Short Version of the International Depression Symptom Scale (IDSS) is comprised of 15 scored items (additional items are assessed for clinical relevance but not included in scoring) assessing symptoms of depression, anxiety, and post-traumatic stress. Each item assesses frequency of experiencing the symptom over the past two weeks, ranging from none of the time (0) to all of the time (3). The IDSS is scored by taking the mean of all items to generate a continuous distress score ranging from 0-3, with higher scores indicating greater distress.
Disease management self-efficacy | Baseline, Endline, Past two weeks
  Disease management self-efficacy will be assessed using a 9-item scale measuring self-reported confidence in taking various actions to manage one's illness, ranging from not confident at all (0) to fully confident (3). Scores will be calculated by taking the mean of all items to generate a continuous score ranging from 0-3, with higher scores indicating greater self-efficacy in managing chronic disease.
Non hypertensive blood pressure | Baseline, Endline, present
  Proportion of individuals who do not have hypertension among the subsample who were hypertensive. Higher proportion is better. Both systolic and diastolic blood pressures will be used.
HbA1C change | Baseline, endline, present
  Proportion of those who could control gluclose in red blood cell (A1C < 6.5) between intervention and control groups. Higher proportion is better. For diabetic subsample
Fasting plasma glucose | Baseline, endline, present.
  Proportion difference of those who could control fasting plasma glucose (FPG<120) of those who could control glucose in red blood cell (AIC<6.5) between intervnetion and comparison gropu. Higher proportion is better. For diabetic subsample
Incidence of seizure | Baseline, Endline, present.
  For epileptic patients, incidence rate ratio of seizures between intervention and comparison groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Mae La Refugee Camp, Mae Sot, Thailand

IPD SHARING:
Plan to Share IPD: No